CLINICAL TRIAL: NCT04976803
Title: A Tissue Collection Study to Explore the Correlation Between ATM Genetic Alterations by Next-Generation Sequencing and ATM Loss-of-Protein Via IHC (ATR-ID Study)
Brief Title: Tissue Collection for Correlation Between ATM Alterations by Next-Generation Sequencing and ATM Loss-of-Protein
Acronym: ATM
Status: Completed | Type: Observational
Sponsor: Artios Pharma Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: ART0380C002
Record Dates: First submitted 2021-07-05; First posted 2021-07-26 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Solid Tumor, Unspecified, Adult
Keywords: ATM; DDR; ATR; protein expression; LoF

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A formalin-fixed tumor tissue block or 5 freshly cut air-dried sections mounted on positively charged slides. Tissue sections cut from the blocks should be 4-5 micron thickness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Deceased patients with archival tissue
  Interventions: Other: Determination of ATM alteration status.
- Group B: Living patients with archival tissue
  Interventions: Other: Determination of ATM alteration status.
- Group C: Living patients without archival tissue
  Interventions: Other: Determination of ATM alteration status.

INTERVENTIONS:
Other: Determination of ATM alteration status. — ATM alterations identified using NGS profiles with ATM protein expression levels from tumor tissue assessed by IHC.

SUMMARY:
This study examines the correlation between ATM alterations identified using NGS profiles with ATM protein expression levels from tumor tissue assessed by IHC.

DETAILED DESCRIPTION:
The purpose of this study is to address whether ATM genomic aberrations could be used to enrich for patients with ATM LoP. Screening of unselected patient populations for ATM protein loss is likely to a lead to high failure rate by IHC testing, as the prevalence of this is expected to be low. This study could allow for identification of the types of ATM aberrations that lead to ATM LoP, and thus significantly decrease IHC failure rate by pre-selecting patients harboring such aberrations. In this study the investigator will be collecting archival tumor tissue or fresh tissue which will be assessed for ATM LoP and compared to NGS data. Additionally, patients whose tumors exhibit ATM LoP within this study could potentially enroll onto the treatment study REFMAL 721/ART0380C001.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the following criteria in order to be included in the research study:

All patients (Groups A, B, and C) must meet the following criteria:

1. Previous genetic testing of ATM genomic aberrations.
2. ≥18 years of age.

   All living patients (Groups B and C) must also meet the additional criteria:
3. Signed written informed consent to access archival tissue, if available.

   All Group C patients must also meet the additional criteria:
4. Provided signed written informed consent to collect a fresh core biopsy.
5. Have a non-irradiated, biopsiable tumor site to allow sampling for analysis via IHC for loss of ATM protein.
6. Potentially eligible for REFMAL 721/ART0380C001:

   * Have not received a previous treatment targeting the ATR/CHK1 pathway.
   * If patients have a germline BRCA mutation or a cancer with a somatic BRCA mutation or which is HRD positive and for which there is an approved PARP inhibitor, patients should have received such treatment.
   * Have an estimated life expectancy of ≥12 weeks, in the judgment of the investigator
   * Advanced or metastatic cancer which is refractory to standard therapies, or for which no standard therapies exist, or for which the investigator feels no other active therapy is required for the duration of the study.
   * Performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) scale

Exclusion Criteria:

There are no exclusion criteria for patients in Group A and Group B.

Group C patients who meet any of the following criteria will be excluded from study entry:

1. Have a significant bleeding disorder or vasculitis or had a Grade 3 bleeding episode within 12 weeks prior to enrollment.
2. Presumed ineligible for enrollment to REFMAL 721/ART0380C001:

   * Psychological, familial, sociological, or geographical conditions that that would compromise the patient's ability to adhere to future procedures likely in a Phase I protocol (such as REFMAL 721/ ART0380C001).
   * Women who are pregnant, breast feeding, or who plan to become pregnant within the next 6 months.
   * Men who plan to father a child within the next 6 months.
   * Have a serious concomitant systemic disorder that would compromise the patient's ability to adhere to a future protocol (REFMAL 721/ ART0380C001) including:

     1. One or more opportunistic HIV/AIDs-related infections within the past 12 months.
     2. Documented active or chronic infection with hepatitis B virus (positive hepatitis B surface antigen [+HBsAg]), or hepatitis C virus.
     3. Known history of clinical diagnosis of tuberculosis.
     4. Have had a malignancy prior to the current malignancy. Patients with carcinoma in situ of any origin and patients with prior malignancies who are in remission and whose likelihood of recurrence is very low (such as basal cell carcinoma), as judged by the medical monitor, are eligible for this study.
   * Have evidence of interstitial lung disease or pneumonitis (whether symptomatic or asymptomatic).
   * Have moderate or severe cardiovascular disease, such as the following:

     1. Have the presence of cardiac disease.
     2. Have valvulopathy that is severe, moderate, or deemed clinically significant.
     3. Have documented major electrocardiogram (ECG) abnormalities which are clinically significant.
   * Have symptomatic or uncontrolled brain metastases, spinal cord compression, or leptomeningeal disease requiring concurrent treatment, including but not limited to surgery, radiation, and/or corticosteroids (patients receiving anticonvulsants are eligible).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with identified ATM alterations will be potentially enrolled into this study in 1 of 3 patient populations
  * Group A: Deceased patients with archival tumor tissue
  * Group B: Living patients with archival tumor tissue
  * Group C: Living patients without archival tumor tissue
Sampling Method: Non-Probability Sample
Enrollment: 229 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with loss of ATM protein | 12 months
  ATM protein expression levels from tumor tissue assessed by immunohistochemistry (IHC)

SECONDARY OUTCOMES:
Number of potential patients with loss of ATM protein eligible for study REFMAL 721/ART0380C001 | 12 months
  Patients in Group C are considered for enrolment into study REFMAL 721/ART0380C001 and must meet eligibility based on review of their medical records. REFMAL 721/ART0380C001 is a phase I/IIa open-label trial to assess the safety, tolerability, and preliminary efficacy of the ATR kinase inhibitor, ART0380 administered as a monotherapy as well as in drug combinations with gemcitabine in patients with advanced or metastatic solid tumors.
Number of ATM genomic aberrations that lead to ATM LoP | 12 months
  Identify types of ATM protein expression from tumor tissue assessed by immunohistochemistry (IHC)
Rate of loss of function (LoF) of the ATM gene in patients with genomic aberrations in the ATM gene | 12 months
  ATM alterations identified using Next-Generation Sequencing(NGS) profiles

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Johnson, MD, Study Chair — Sarah Cannon
Locations (3):
- United States (2):
  - Oklahoma University, Oklahoma City, Oklahoma
  - Tennessee Oncology, Nashville, Tennessee
- Sarah Cannon Research UK, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No